CLINICAL TRIAL: NCT06601894
Title: The Relationship of Platelet Counts With Sickle Cell Anemia in the Eastern Region of Saudi Arabia
Status: Not yet recruiting | Type: Observational
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Khalid Ali Majrashi, Student, Majmaah University
Other Study IDs: IRB Log No.: 29-EP-2024
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Anaemia; SCD
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Males: The study will be conducted on CBC count special PLT for adult Males of different ages with sickle cell anemia.
  Interventions: Diagnostic Test: Platelets count
- Children: The study will be conducted on CBC count special PLT for adult Males of different ages with sickle cell anemia.
  Interventions: Diagnostic Test: Platelets count
- Females: The study will be conducted on CBC count special PLT for adult Males of different ages with sickle cell anemia.
  Interventions: Diagnostic Test: Platelets count

INTERVENTIONS:
Diagnostic Test: Platelets count — the study include will take medical investigation data for all sickle cell patients.

SUMMARY:
This study aims to evaluate the relationship between platelet counts and sickle cell disease in the eastern region of the Kingdom of Saudi Arabia.

DETAILED DESCRIPTION:
Introduction:

This study aims to evaluate the relationship between platelet counts and sickle cell disease in the eastern region of the Kingdom of Saudi Arabia.

Purpose: This study aims to assess the prevalence and factors associated with elevated platelet counts in people with sickle cell disease in the eastern region of Saudi Arabia.

Methods: This cross-sectional study at Majmaah University will analyze prerecorded data frfom the eastern region of Saudi Arabia to investigate the relationship between platelet counts and sickle cell disease, identifying associated factors and assessing the link .

Importance: To assess the relationship between platelet counts and disease severity in Pationt with SCD.

Aim :To investigate the relationship between platelet counts and SCD in the eastern region of the Kingdom of Saudi Arabia.

ELIGIBILITY:
Inclusion criteria: All the diagnosed patients of sickle cell disease regardless of age and gender.

Exclusion criteria: Patients without having sickle cell disease regardless of age and gender.

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include a cohort of people with SCD who are registered at the Hereditary Blood center al-ahssa.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Collecting platelet data for sickle cell anemia patients | From January 2023 to December 2023
  Collecting platelet data for sickle cell anemia patients in males and female and children based on different ages, then analyzing them and studying their relationship

CONTACTS AND LOCATIONS:
Overall Officials: Khalid A Majrashi, Principal Investigator — Majmaah University
Locations (1):
- Khalid Ali Majrashi, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wun T, Paglieroni T, Rangaswami A, Franklin PH, Welborn J, Cheung A, Tablin F. Platelet activation in patients with sickle cell disease. Br J Haematol. 1998 Mar;100(4):741-9. doi: 10.1046/j.1365-2141.1998.00627.x. PMID 9531343
- [Result] Shome DK, Jaradat A, Mahozi AI, Sinan AS, Ebrahim A, Alrahim M, Ebraheem MS, Mansoor EJ, Majed KS, Azeez Pasha SA. The Platelet Count and its Implications in Sickle Cell Disease Patients Admitted for Intensive Care. Indian J Crit Care Med. 2018 Aug;22(8):585-590. doi: 10.4103/ijccm.IJCCM_49_18. PMID 30186009
- [Result] Yee MEM, Batsuli G, Chonat S, Park S. Thrombocytosis with acquired von Willebrand disease in an adolescent with sickle cell disease. Clin Case Rep. 2020 Nov 20;9(1):457-460. doi: 10.1002/ccr3.3556. eCollection 2021 Jan. PMID 33489197